CLINICAL TRIAL: NCT01462123
Title: Resect and Discard Strategy in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Valduce Hospital (Other)
Other Study IDs: RD 2010
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Endoscopic Assessment; Colonic Polyps; Endoscopic Surveillance; NBI
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- small polyps patients: Patients with one small polyps at colonoscopy
  Interventions: Other: endoscopic assessment of colonic polyps

INTERVENTIONS:
Other: endoscopic assessment of colonic polyps

SUMMARY:
Nowadays, post-polypectomy surveillance intervals are determined by combining endoscopic and pathologic data. Real-time imaging technologies, have shown promising results in discriminating adenomatous from non-adenomatous polyps.

The "resect and discard strategy" for small polyps (based on real-time assessment of the histology and on the endoscopic resection without pathological examination) has been shown to be cost-effective in simulation models. No data exist about the impact of this strategy in clinical practice.

The aim of present study was to assess whether the systematic use, in the everyday clinical practice, of the "resect and discard strategy" allows to correctly manage patients with small colonic polyps.

ELIGIBILITY:
Inclusion Criteria:

* consecutive adult outpatients undergoing colonoscopy for routine clinical indications

Exclusion Criteria:

* surveillance interval was not necessarily directed by endoscopic findings (history of colorectal cancer, inflammatory bowel disease, hereditary polyposis syndromes, hereditary non-polyposis colorectal cancer)
* colonoscopy was performed without NBI technology
* at least one lesion > 10 mm or < 10 mm but with morphologic features suspect for malignancy (depressed or ulcerated lesions) was detected
* bowel preparation was inadequate
* caecal intubation was not accomplished
* polyps could not be resected for concomitant anticoagulation treatment, 7) polyps were resected but not retrieved for pathology.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult outpatients undergoing colonoscopy for routine clinical indications
Sampling Method: Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2011-02

PRIMARY OUTCOMES:
The primary outcome of the study was to assess the agreement between "endoscopy-" and "histology-determined" surveillance strategies after small adenoma resection.

SECONDARY OUTCOMES:
sensitivity of the endoscopic assessment (WL coupled with NBI) of small (<10 mm) adenomas
operative characteristics for the diagnosis of diminutive (< 5 mm) adenomas
the feasibility of non histologic evaluation, represented by the proportion of polyps in which a in-vivo diagnosis of adenoma can be made with high confidence
specificity of the endoscopic assessment
accuracy of the endoscopic assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Valduce Hospital - Gastroenterology Department, Como, CO, Italy

REFERENCES:
- [Derived] Paggi S, Rondonotti E, Amato A, Terruzzi V, Imperiali G, Mandelli G, Terreni N, Lenoci N, Spinzi G, Radaelli F. Resect and discard strategy in clinical practice: a prospective cohort study. Endoscopy. 2012 Oct;44(10):899-904. doi: 10.1055/s-0032-1309891. Epub 2012 Aug 2. PMID 22859259